CLINICAL TRIAL: NCT04210089
Title: Total Contact Soft Cast in Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORSU-2019-28102
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer; Diabetes Mellitus; Foot Ulcer; Foot Ulcer, Diabetic; Ulcer; Ulcer Foot; Ulcer, Leg; Ankle Ulcer
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer; Ulcer; Leg Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Soft Cast with a Removable Cam Boot (Experimental): Patients with a foot, ankle, or lower leg ulcer (which we expect to be mostly diabetic foot ulcers) will be provided with a total contact soft cast with removable cam boot.
  Interventions: Device: Total Contact Soft Cast; Device: Cam Boot
- Soft Cast without a Removable Cam Boot (Experimental): Patients with a foot, ankle, or lower leg ulcer (which we expect to be mostly diabetic foot ulcers) will be provided with a total contact soft cast.
  Interventions: Device: Total Contact Soft Cast
- Conventional (No Intervention): Patients with a foot, ankle, or lower leg ulcer (which we expect to be mostly diabetic foot ulcers) will use conventional offloading including total contact casting, removable cast boots (cam boots), CROW boots, bracing, AFO's, offloading shoes, insoles, padding, shoe modifications, crutches, wheelchairs, rollabout, and surgical correction.

INTERVENTIONS:
Device: Total Contact Soft Cast — The total contact soft cast will consist of wound dressing of choice to the ulcer and a plantar foot accommodative offloading felt pad for all foot ulcers, with 4x4 gauze pads added to the arch to create a rocker bottom for metarsophalangeal joint (MPJj) and plantar heel ulcers. The next layers will be:
  * Unna boot from MPJs to just below the knee,
  * Sterile Kerlix from MPJs to just below the knee
  * Sterile 4 inch Kling wrap from the MPJs to just below the knee,
  * Four inch coban from MPJs to just below the knee, and
  * Ace wraps from MPJs to just below the knee
  Arms: Soft Cast with a Removable Cam Boot; Soft Cast without a Removable Cam Boot
Device: Cam Boot — Removable Diabetic cam boot will be used in patients willing and capable of using it. If patient does not want to use Diabetic cam boot then surgical shoe or regular shoe would be options.
  Arms: Soft Cast with a Removable Cam Boot

SUMMARY:
To determine the effectiveness, compliance, patient tolerance, ease of use and safety of total contact soft cast in diabetic foot ulcers.

DETAILED DESCRIPTION:
This study will evaluate whether the use of a total contact soft cast with or without a removable cam boot is as effective in healing diabetic foot ulcers as more commonly used offloading methods.

The total contact soft cast will consist of wound dressing of choice to the ulcer and a plantar foot accommodative offloading felt pad for all foot ulcers, with 4x4 gauze pads added to the arch to create a rocker bottom for metarsophalangeal joint (MPJj) and plantar heel ulcers. The next layers will be:

* Unna boot from MPJs to just below the knee,
* Sterile Kerlix from MPJs to just below the knee
* Sterile 4 inch Kling wrap from the MPJs to just below the knee,
* Four inch coban from MPJs to just below the knee, and
* Ace wraps from MPJs to just below the knee

Removable diabetic cam boot will be used in patients willing and capable of using it. If patient does not want to use diabetic cam boot then surgical shoe or regular shoe would be options.

ELIGIBILITY:
Inclusion Criteria:

- Any adult with a diabetic foot ulcer

Exclusion Criteria:

* Allergy to Calamine or Zinc oxide
* Inability to have leg wrapped
* Inability to be seen weekly or as needed
* Unable or unwilling to consent
* Prisoners
* Persons lacking capacity to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete Healing Rates | 16 weeks
  Complete healing is defined as complete epithelization of the ulcer. Outcome will be reported in days.

SECONDARY OUTCOMES:
Patient Compliance with Use of the Total Contact Soft Cast | 16 weeks
  The percentage of patients who use the total contact soft cast until complete healing or 16 weeks of treatment will be calculated.
Patient Complications | 16 weeks
  The percentage of patients who need to stop using the soft case due to complications will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Schuster, DPM, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No